CLINICAL TRIAL: NCT01543997
Title: Investigating Clinical Benefits of a Novel Sleep-focused Mind-body Program on Gulf War Illness (GWI) Symptoms: An Exploratory Randomized Controlled Trial
Brief Title: Clinical Benefits of a Novel Sleep-focused Mind-body Program on Gulf War Illness (GWI) Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: VA Salt Lake City Health Care System (U.S. Federal Agency); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Yoshio Nakamura, Research Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00049003
Record Dates: First submitted 2012-02-27; First posted 2012-03-05 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Sleep Disturbance; Persian Gulf War Syndrome in Veteran
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mind-Body Bridging Program (Experimental): The Mind-Body Bridging Program (MBBP) is an awareness training program (ATP)to help individuals improve their health condition and attain a state of well-being. Bridging is the primary technique that facilitates the healing process, by bringing one back to the present moment to experience thoughts, emotions and physical sensations. Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Interventions: Behavioral: Mind-Body Bridging Program
- Supportive Education (Active Comparator): Supportive Education program will provide educational lectures on disability, sleep hygiene, and current research on depression and non-directive, supportive discussions about these topics.
  Interventions: Behavioral: Supportive Education

INTERVENTIONS:
Behavioral: Mind-Body Bridging Program — Bridging aims to reduce the impact of negative thought patterns that contribute to stress in the body.
  Other Names: MBBP
  Arms: Mind-Body Bridging Program
Behavioral: Supportive Education — This intervention will provide educational lectures on disability, sleep hygiene, and current research on depression and nondirective, supportive discussions about these topics.
  Other Names: SED
  Arms: Supportive Education

SUMMARY:
The purpose of this study is to investigate clinical benefits of a novel sleep-focused mind-body program on Gulf War Illness (GWI) symptoms.

DETAILED DESCRIPTION:
This randomized study investigates whether two treatment conditions:Mind-Body Bridging (MBB) and Supportive Education (SED) are effective in improving sleep disturbance and self-reported indicators of other co-morbid symptoms in veterans with GWI. The two treatment conditions will each comprise 3 sessions of 2 hr. duration and conducted over 3 consecutive weeks (Week 1-3).

ELIGIBILITY:
Inclusion Criteria:

* Veteran from First Gulf War
* Suffering from sleep disturbance
* Has other chronic symptoms of Gulf War Illness:

  * fatigue
  * chronic headaches
  * joint/muscle pain
  * cognitive difficulties
  * memory/concentration problems
  * shortness of breath
  * gastrointestinal symptoms

Exclusion Criteria:

* terminally ill
* a highly unstable medical or psychiatric condition
* Parkinson disease
* dementia of any cause
* Nocturia
* delayed/advanced sleep phase syndrome
* Narcolepsy

Ages: 38 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-01; Primary Completion 2015-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the measure of the Medical Outcomes Study-Sleep Scale | Week1, Week2, Week 3, Week 4, Week 15
Change from baseline in the measure of the Sleep Diary | Week2, Week 4, Week 15

SECONDARY OUTCOMES:
Pain | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  Multidimensional Pain Inventory Pain Scale
Fatigue | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  Multidimensional Fatigue Inventory
Cognitive functioning | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  Cognitive Failures Questionnaire
Mindfulness | Pre (Baseline), Weekly for 3 weeks, Post (Week4), Follow-up (Week 15)
  5-factor M questionnaire
Health-related quality of life | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  Medical Outcomes Study Short Form-36
PTSD | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  PTSD Check List-Military (PCL-M)
Depression | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  Center of Epidemiological Study-Depression Scale
Psychological symptoms | Pre (Baseline), Post (Week4), Follow-up (Week 15)
  Brief Symptom Inventory 18

CONTACTS AND LOCATIONS:
Overall Officials: Yoshio Nakamura, Ph.D., Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - Pain Research Center, Salt Lake City, Utah
  - VA SLC Health Care System, Salt Lake City, Utah

REFERENCES:
- [Derived] Nakamura Y, Lipschitz DL, Donaldson GW, Kida Y, Williams SL, Landward R, Glover DW, West G, Tuteja AK. Investigating Clinical Benefits of a Novel Sleep-Focused Mind-Body Program on Gulf War Illness Symptoms: A Randomized Controlled Trial. Psychosom Med. 2017 Jul/Aug;79(6):706-718. doi: 10.1097/PSY.0000000000000469. PMID 28406803